CLINICAL TRIAL: NCT02396329
Title: Chlorhexidine Versus Povidone-iodine Antisepsis for Reduction of Post Cesarean Section Surgical Site Infection Rate:a Randomized Controlled Trial
Brief Title: Chlorhexidine Versus Povidone-Iodine Antisepsis for Reduction of Post Cesarean Section Surgical Site Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AMR HELMY YEHIA, MD,MRCOG, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: antisepsis 1
Record Dates: First submitted 2015-03-01; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Chlorhexidine; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chlorhexidine _based antisepsis (Experimental): Including cases undergoing elective&non elective caesarean section.Patients will be were prepared similarly by three applications of 2%chlorhexidine solution time given between each application about 30 seconds followed by drying with a sterile towel and three applications of 70% alcohol after one minute The area scrubbed was from the xiphoid to the knee, reaching the midaxillary line laterally. In both groups, patients received preoperative prophylactic i.v antibiotics (cefotrixone 1 gm) one hour before skin incision.
  .
  Interventions: Drug: Chlorhexidine
- povidone_iodine based antisepsis (Active Comparator): Including cases undergoing elective&nonelective caesarean section.Patients will be scrubbed preoperative with an applicator that contain 10%povidone-iodine scrub aqueous solution(3 consecutive applications)followed by drying with sterile towel and 3 application of 70% alcohol after one minute The area scrubbed was from the xiphoid to the knee, reaching the midaxillary line laterally. In both groups, patients received preoperative prophylactic i.v antibiotics (cefotrixone 1 gm) one hour before skin incision
  Interventions: Drug: Povidone-Iodine

INTERVENTIONS:
Drug: Chlorhexidine
  Arms: chlorhexidine _based antisepsis
Drug: Povidone-Iodine
  Other Names: Betadine
  Arms: povidone_iodine based antisepsis

SUMMARY:
There is no difference between using chlorhexidine-based antisepsis protocol versus povidone-iodine protocol in reduction of surgical site infection in women undergoing cesarean section.

DETAILED DESCRIPTION:
The aim of this study is to examine the efficacy &safety of Chlorhexidine-based antisepsis protocol versus povidone- iodine protocol used as preoperative skin antisepsis for patients undergoing cesarean section in reduction of surgical site infection.Chlorhexidine is a chemical antiseptic. It is effective on both Gram-positive and Gram-negative bacteria, although it is less effective with some Gram-negative bacteria. It has both bactericidal and bacteriostatic mechanisms of action, the mechanism of action being membrane disruption.

Iodine is commonly used as an antiseptic agent clinically. Iodine is usually formulated as an iodophor, which consists of iodine combined with a carrier molecule. This formulation increases the solubility of iodine and provides a reservoir for sustained release. The most commonly used iodophor is povidone iodine which is a 10% iodophor solution that contains 1% available iodine. Iodine molecules penetrate microbial cell walls and cause oxidation of cysteine, iodination of amino acids and unsaturated fatty acids. This leads to reduced protein synthesis and bacterial cell wall damage.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years of age or older who will undergo cesarean deliveries who are at term (37wks-41wks of gestation).
2. Body mass index (BMI) between 20-35kg/m2.
3. Able to communicate well with the investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Rupture of membranes.
2. Patients who have history of allergy to chlorhexidine, alcohol and iodophors.
3. Documented concomitant infections like: Chorioamnionitis, Pyelonephritis, Urinary tract infection, Mastitis.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 410 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection within one week after surgery | One week

SECONDARY OUTCOMES:
Surgical site infection within 30 days after surgery | in 30 days
Long hospital stay | 30 days
  hospital admission for more than 5 days
Hospital readmission | 30 days
  readmission due to sepsis
Febrile morbidity | 10 days
  an oral temperature of 38.0 degree Celsius)or more on any two of the first 10 days postpartum, exclusive of the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: AMR YEHIA, MD, MRCOG, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Hadiati DR, Hakimi M, Nurdiati DS, Masuzawa Y, da Silva Lopes K, Ota E. Skin preparation for preventing infection following caesarean section. Cochrane Database Syst Rev. 2020 Jun 25;6(6):CD007462. doi: 10.1002/14651858.CD007462.pub5. PMID 32580252